CLINICAL TRIAL: NCT01516515
Title: A Double-blind, Randomized, Vehicle-controlled, Parallel-group, Phase II Study to Evaluate the Efficacy and Safety of SR-T100 Gel in Patients With Actinic Keratosis (AK)
Brief Title: Efficacy and Safety Phase II Study of SR-T100 to Treat Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GESRTAKB
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; AK
MeSH Terms: conditions — Keratosis, Actinic | interventions — SR-T100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo, gel (Placebo Comparator): placebo comparator
  Interventions: Drug: Vehicle gel
- SR-T100 with 2.3% of SM, gel (Active Comparator): 2.3% of SM in Solanum undatum plant extract
  Interventions: Drug: SR-T100 with 2.3% of SM

INTERVENTIONS:
Drug: Vehicle gel — placebo
  Arms: placebo, gel
Drug: SR-T100 with 2.3% of SM — 2.3% of SM in Solanum undatum plant extract
  Other Names: SR-T100
  Arms: SR-T100 with 2.3% of SM, gel

SUMMARY:
This Phase II study is to evaluate the efficacy of SR-T100 gel with 2.3% of SM in Solanum undatum plant extract in patient with Actinic Keratosis (AK).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; aged ≥ 18 years old.
2. Patient who accepts to enter the study by signing written informed consent.
3. Patient has 4 to 8 clinically diagnosed, discrete, non-hyperkeratotic, non-hypertrophic AK, located with or without a contiguous 25cm2 areas.
4. Patient allows biopsy to be performed on selected lesion.
5. Patient agrees to apply the study medication on prescribed treatment area with an occlusive dressing at least 20 hours per day.
6. Patient agrees photographs to be taken on selected lesion and used as part of the study data package.
7. Patient in good general health condition (performance status ≤ 2 Eastern Cooperative Oncology Group (ECOG).
8. Sexually active female patient with child-bearing potential must take reliable contraception method(s) during the participation of the study.

Exclusion Criteria:

1. Patient with recurrent invasive squamous cell carcinoma (SCC).
2. Patient has grossly suspicious or inflamed lymph nodes on physical examination.
3. Patient has evidence of clinically significant or unstable medical conditions.
4. Patient has any skin condition in the treatment area that may be made worse by treatment.
5. Patient currently uses or had used on the treatment area(s) OTC retinol products, corticosteroids, cryosurgery, curettage, 5-fluorouracil (5-FU), imiquimod, topical diclofenac, retinoids, or other topical AK treatments (such as laser abrasion, dermabrasion, glycolic acids, or chemical peels) 28 days prior to screening visit.
6. Patient had received systemic cancer chemotherapy or immunosuppressant; on the target evaluation area that psoralen plus UVA therapy, UVB therapy were treated 6 months prior to screening visit.
7. Patient currently uses or has used prednisone and/or prednisolone (≥ 10 mg or the equivalent) more than 2 weeks continuously within 12 weeks prior to randomization visit.
8. Engaging in activities involving excessive or prolonged exposure to sunlight.
9. History of allergy or sensitivity to related compounds or other components of the investigational product formulation.
10. Woman who is pregnant, lactating or planning to become pregnant during the study.
11. Patient used any investigational drug within 8 weeks prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-02; Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Total clearance rate: | 8-week post-EOT visit (scheduled at Week 24 visit)
  The proportion of patients achieving total clearance of AK lesions in the treatment area (in total of 25cm2 area) at 8-week post-EOT visit (scheduled at Week 24 visit) .

SECONDARY OUTCOMES:
Partial clearance rate | 24 week
  The proportion of patients achieving ≥ 75% total clinically assessed AK lesion counts out of all target lesions in the treatment area (in total of 25cm2 area) at the post-EOT visit (8 weeks after EOT visit).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Contour Dermatology & Cosmetic Surgery Center, Rancho Mirage, California
  - IMMUNOe International Research Centers, Longmont, Colorado
  - Atlantic Clinical Research Collaborative, West Palm Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Suzanne Bruce and Associates,P.A. The Center for Skin Research, Katy, Texas
  - Pflugerville Dermatology Clinical Research, Pflugerville, Texas
  - The Education & Research Foundation, Inc, Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington